$\frac{\hbox{Title:}}{\hbox{Informed Decisions and Patient Outcomes: An Interdisciplinary Approach to Chronic Hip Pain.}}$ 

NCT03519087

Document dates: 2019.03.20 (Cr (Created)

(Uploaded to clinicaltrials.gov) 2019.09.30

# Data Analysis Plan

Primary outcome measures:

# 1. Treatment plan

Chi-squared test will be used to compare the distribution of participants who included physical therapy in their post-evaluation treatment plan in the interdisciplinary group compared to the standard group ( $P \le 0.05$ ).

## 2. Decisional conflict

A Mann-Whitney U test will be used to compare post-evaluation decisional conflict between the interdisciplinary and standard groups (P<0.05).

Secondary outcome measures:

1. Changes in provider protocol opinions

A single-rater will evaluate qualitative interviews of providers to quantify the number of responses within the following pre-determined themes: implementation, physical therapy evaluation, time, patient response, clinical reasoning, environment.

# 2. Participant protocol opinions

Participants did not participate in qualitative interviews due to resource limitations.

# 3. Decisional conflict (x4 weeks)

Evaluation of any changes in decisional conflict over the 3-week intervention period will be limited by small sample size. Descriptive statistics may be reported for those who received or did not receive posture and movement training.

### 4. Patient-reported hip function (x4 weeks)

Evaluation of any changes in patient-reported hip function over the 3-week intervention period will be limited by small sample size. Descriptive statistics may be reported for those who received or did not receive posture and movement training.

## 5. Movement mechanics

Evaluation of any changes in kinematics or kinetics over the 3-week intervention period will be limited by small sample size. Analysis of these data were not completed due to stoppage of funding and limited personnel.

# 6. Decisional regret

Decisional regret was collected but will not be analyzed due to lack of construct validity.

# 7. Hip strength

Evaluation of any changes in hip strength over the 3-week intervention period will be limited by small sample size. Descriptive statistics may be reported for those who received or did not receive posture and movement training.